CLINICAL TRIAL: NCT04564079
Title: A Multi-Centre Observational Study to Evaluate the Clinical Utility of Returning Genomic Aberration Results Using the Oncomine Precision Assay in Advanced or Metastatic Non-Small Cell Lung Cancer Within the Exactis Network
Brief Title: An Observational Study to Evaluate the Clinical Utility of the Oncomine Precision Assay Within the Exactis Network
Status: Completed | Type: Observational
Sponsor: Exactis Innovation (Other)
Responsible Party: Sponsor
Other Study IDs: Exactis-01
Record Dates: First submitted 2020-08-28; First posted 2020-09-25 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: NSCLC
Keywords: Genomic Aberrations; Exactis Network; Advanced or Metastatic Non-Small Cell Lung Cancer; Liquid Biopsy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples and/or tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A Multi-centre Observational Study to Evaluate the Clinical Utility of Returning Genomic Aberration results Using the Oncomine Precision Assay in Advanced or Metastatic Non-Small Cell Lung Cancer Patients within the Exactis Network

DETAILED DESCRIPTION:
This prospective multi-center observational study will evaluate the clinical utility of returning genomic aberration results in blood and/or tissue using the Oncomine Precision Assay in non-small cell lung cancer (NSCLC) patients. Up to 100 patients with stage IIIb/IV NSCLC will consent to have their blood and tissue profiled on the Oncomine Precision Assay. A baseline plasma sample will be collected for all patients, of which up to 50 patients will have a tissue sample collected from pathology archives or planned biopsy or surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with NSCLC, which is (i) advanced or metastatic (stage IIIb/IV), (ii) non- squamous histology NSCLC as confirmed by local histopathology (mixed squamous and adenocarcinoma is allowed), and has (iii) radiographically measurable disease with at least one bidimensionally measurable lesion of > 1 cm by CT scan
* No prior treatment for advanced or metastatic NSCLC, except for palliative radiation therapy to non-lung or non-thorax metastases. Patients who received palliative radiation therapy to metastases located within or approximately to the lung or thorax must be evaluated for eligibility.
* Willing and able to provide adequate blood sample prior to starting treatment.
* Willing to provide primary or metastatic tissue, if available.
* Signed and dated Research Ethics Board (REB)-approved informed consent form for Exactis-01 or PMT.
* Not pregnant or breastfeeding

Exclusion Criteria:

• Patients who have a history of another active cancer within the past 2 years from date of consent except cervical cancer in situ, basal cell carcinoma of the skin or another in situ carcinoma that is considered cured by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with NSCLC, which is i) advanced or metastatic (stage IIIb/IV), ii) non-squamous histology NSCLC as confirmed by local histopathology (mixed squamous and adenocarcinoma is allowed).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
To compare the number of genomic aberrations detected by the Oncomine Precision Assay vs Standard of Care | 1 year
  Proportion of patients for whom an actionable genomic aberration is detected in at least one of the eight genes (ROS1, ERBB2, MET, BRAF, KRAS, RET, ALK, EGFR) using the Oncomine Precision Assay vs. study site's standard of care

SECONDARY OUTCOMES:
Clinical utility of returning genomic aberration results by quantifying the number of patients who received targeted therapy based on results returned from the Oncomine Precision Assay genomic aberration results in blood and/or tissue | 2 years
Clinical utility of returning genomic aberration results by quantifying the number of patients enrolled on a clinical trial based on results returned from the Oncomine Precision Assay in blood and/or tissue | 2 years

OTHER OUTCOMES:
Exploratory - Analytical validity of Oncomine Precision Assay | 2 years
  Number of genomic aberrations concordant and discordant between tissue and blood using the Oncomine Precision Assay
Exploratory- Sensitivity and specificity of mutation detection analysis of extracellular vesicles (EV) total nucleic acids | 2 years
  Compare the sensitivity and specificity of mutation detection in extracellular vesicles (EV) total nucleic acids and circulating tumor total nucleic acids
Exploratory- Explore the response patterns to treatment based on EV RNAs | 2 years
  Small RNA extracted from plasma EV at baseline and at progression will be analyzed using RNA sequencing. Potential association between expression profiles and clinical parameters such as treatment response will be explored and candidate patterns predictive of treatment response will be tested using artificial intelligence algorithms.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Agulnik, MD, Principal Investigator — Principal Investigator
Locations (6):
- Canada (6):
  - Centre hospitalier universitaire Dr-Georges-L.-Dumont, Moncton, New Brunswick
  - The Moncton Hospital, Moncton, New Brunswick
  - The Ottawa Hospital, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - Centre hospitalier universitaire de Sherbrooke (CHUS), Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Yes
As in the PMT registry, data and samples will be collected, coded and stored in secure and protected installations. Information and samples provided to researchers will be double-coded so that they cannot be traced back to you. Exactis takes great care to protect participants' data and samples, to minimize security risks and the possibility of a confidentiality breach.

REFERENCES:
- See also: exactis.ca — https://www.exactis.ca
- See also: PMT registry — http://clinicaltrials.gov/ct2/show/NCT02355171?term=personalize+me+treatment&draw=2&rank=9